CLINICAL TRIAL: NCT05071794
Title: Effect of Propofol on Postoperative Nausea and Vomiting in Patients Undergoing Elective Cesarean Section Under Spinal Anesthesia.
Brief Title: Effect of Propofol on Postoperative Nausea and Vomiting.
Acronym: (PONV)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pakistan Air Force (PAF) Hospital Islamabad (Other)
Responsible Party: Principal Investigator, Atif Nazir, Registrar Anesthesiologist, Pakistan Air Force (PAF) Hospital Islamabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PAFHIslamabad
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: postoperative nausea and vomiting, propofol
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting | interventions — Propofol; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): Subhypnotic dose of propofol, 0.5mg/kg, 10 - 15 min before end of surgery
  Interventions: Drug: Propofol
- Placebo (Placebo Comparator): Normal saline 0.9%, 10 mL , 10 - 15 min before end of surgery
  Interventions: Drug: saline 0.9%

INTERVENTIONS:
Drug: Propofol — Antiemetic effect of propofol
  Other Names: propofol injection
  Arms: Propofol
Drug: saline 0.9% — Placebo
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
As PONV is an unpleasant experience that badly affects the patients' quality of life after surgery and the anti-emetic effects of propofol have been seldomly studied in Pakistan, this study aims at investigation of the beneficial effects of propofol in reducing the occurrence of PONV.

DETAILED DESCRIPTION:
Cesarean Section is one of the most commonly performed surgical procedures in the obstetric patients. Adequate intra and postoperative analgesia is very important in providing comfort to the mother, early breastfeeding, ambulation and discharge as well as enhancing patient satisfaction.Spinal anesthesia is widely accepted as the anesthesia of choice for cesarean section owing to its safety and speed. PONV is an unpleasant condition, often underestimated side effect of anesthesia and surgery, quite common in women undergoing spinal anesthesia for cesarean.It is one of the significant problems in Post Anaesthesia Care Units. The etiology of PONV is multifactorial with patient factors (gender, history of motion sickness, age), intra Op factors (type of anesthesia, surgery and opioid use) and post Op factors (pain, post Op opioid use) which are found to be associated with the PONV. Apfel simplified scoring is based on four independent factors including female gender, non-smoker, history of PONV or motion sickness and use of opioids. Each predictor is given a score of 1. A score of 0,1,2,3 or 4 predicts the chance of developing PONV as approximately 10%, 20%, 40% or 80%.

The intense efforts accompanying emesis increase the risk of complications such as wound dehiscence, bleeding, aspiration pneumonitis, dehydration, electrolyte imbalance and interference with nutrition. While it is difficult to completely avoid the occurrence of PONV, it can be markedly reduced using a multimodal non-opioid analgesia, total intravenous anesthesia and adequate prophylactic antiemetic premedication. Propofol has been reported to have anti-emetic effects at sub hypnotic dose as a bolus or a continuous infusion in susceptible individuals undergoing surgeries, though the exact mechanism of this effect is yet to be discovered.

In a research published in BMC Anesthesiology, the data indicates a significant difference in the incidence of PONV in control group (93.9%) and the study group (8.7%) with a single sub hypnotic dose of propofol administered 10-15 min before the end of surgery in parturients undergoing cesarean section under spinal anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Parturient aged between 18 - 50 years
* Elective Cesarean under spinal anesthesia
* Patients at increased risk of PONV based on Apfel score 2 or more
* ASA Class II
* Ability to give informed consent

Exclusion Criteria:

* Allergy to propofol
* ASA Class III and above
* Anti emetic drug administered 24 hrs prior to surgery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2022-10-29 (Actual)

PRIMARY OUTCOMES:
postoperative nausea and vomiting | 1 hour stay in Postanaesthesia Care Unit
  Subjective complaint of nausea or any episode of vomiting

CONTACTS AND LOCATIONS:
Overall Officials: ATIF NAZIR, MD, Principal Investigator — PAF Hospital Islamabad
Locations (1):
- PAF Hospital Islamabad, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niu K, Liu H, Chen RW, Fang QW, Wen H, Guo SM, Williams JP, An JX. Use of propofol for prevention of post-delivery nausea during cesarean section: a double-blind, randomized, placebo-controlled trial. J Anesth. 2018 Oct;32(5):748-755. doi: 10.1007/s00540-018-2549-x. Epub 2018 Sep 12. PMID 30209576
- [Background] Shaikh SI, Nagarekha D, Hegade G, Marutheesh M. Postoperative nausea and vomiting: A simple yet complex problem. Anesth Essays Res. 2016 Sep-Dec;10(3):388-396. doi: 10.4103/0259-1162.179310. PMID 27746521
- [Background] Urits I, Orhurhu V, Jones MR, Adamian L, Borchart M, Galasso A, Viswanath O. Postoperative Nausea and Vomiting in Paediatric Anaesthesia. Turk J Anaesthesiol Reanim. 2020 Apr;48(2):88-95. doi: 10.5152/TJAR.2019.67503. Epub 2019 Nov 11. PMID 32259138
- [Background] Kim EG, Park HJ, Kang H, Choi J, Lee HJ. Antiemetic effect of propofol administered at the end of surgery in laparoscopic assisted vaginal hysterectomy. Korean J Anesthesiol. 2014 Mar;66(3):210-5. doi: 10.4097/kjae.2014.66.3.210. Epub 2014 Mar 28. PMID 24729843
- [Background] Jelting Y, Klein C, Harlander T, Eberhart L, Roewer N, Kranke P. Preventing nausea and vomiting in women undergoing regional anesthesia for cesarean section: challenges and solutions. Local Reg Anesth. 2017 Aug 9;10:83-90. doi: 10.2147/LRA.S111459. eCollection 2017. PMID 28860857
- [Result] Kampo S, Afful AP, Mohammed S, Ntim M, Buunaaim ADB, Anabah TW. Sub-hypnotic dose of propofol as antiemetic prophylaxis attenuates intrathecal morphine-induced postoperative nausea and vomiting, and pruritus in parturient undergoing cesarean section - a randomized control trial. BMC Anesthesiol. 2019 Sep 14;19(1):177. doi: 10.1186/s12871-019-0847-y. PMID 31521119